CLINICAL TRIAL: NCT02851368
Title: A Pilot Trial of Near Infrared Fluorescence Imaging With Indocyanine Green in the Detection and Diagnosis of Neoplastic Pulmonary Nodules
Brief Title: Near Infrared Fluorescence Imaging With Indocyanine Green
Acronym: NIFI-ICG
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Inderpal Sarkaria, MD, MD, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCI 15-205
Record Dates: First submitted 2016-07-05; First posted 2016-08-01 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Solitary Pulmonary Nodules
Keywords: Indocyanine Green; Fluorescence Imaging
MeSH Terms: conditions — Solitary Pulmonary Nodule | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Near Infrared Fluorescence Imaging with Indocyanine Green (Other): Patients will receive an injection of indocyanine green (ICG) 1 day prior to surgery. Near infrared fluorescence imaging (NIFI) will be used to identify pulmonary nodules during the surgical biopsy and/or resection procedure.
  Interventions: Device: near infrared fluorescence imaging (NIFI); Drug: Indocyanine Green

INTERVENTIONS:
Device: near infrared fluorescence imaging (NIFI) — The NIFI system will be evaluated for its ability to 1) visualize nodules and their margins 2) differentiate between benign and malignant nodules and 3) identify additional undiagnosed nodules after receiving an injection of indocyanine green 1 day prior to planned surgery.
Drug: Indocyanine Green — Indocyanine Green will be administered intravenously 1 day prior to NIFI.

SUMMARY:
This research study will evaluate how Near Infrared Fluorescence imaging (NIFI) with indocyanine green (ICG) contrast dye can assist in the identification and diagnosis of lung nodules during surgery. NIFI is an intraoperative imaging technology that utilizes a coupled camera/fluorophore (ICG) system to fluoresce tissues of interest. Intravenous ICG is a fluorophore with a long-standing high safety profile.

DETAILED DESCRIPTION:
This research study is a pilot test of the effectiveness of a near infrared fluorescence imaging (NIFI) system in the detection and diagnosis of pulmonary nodules. Patients selected for enrollment in this study will be adults (≥18 years) that have been scheduled for surgical biopsy and/or resection of a primary lung nodule identified by prior imaging. Patients will receive an injection of indocyanine green (ICG) contrast dye one day prior to their surgery. Intraoperatively, the NIFI system will be used to visualize and characterize the fluorescence patterns given off by these lung nodules, as well as look for additional undiagnosed nodules. These nodules will then be resected and receive histological characterization, as per standard of care. The NIFI system will be evaluated for its ability to 1) visualize nodules and their margins 2) differentiate between benign and malignant nodules and 3) identify additional undiagnosed nodules.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing to undergo surgical biopsy and/or resection of pulmonary nodule(s).
* Women and men at least 18 years of age
* Subjects must have a CT scan of the chest within 8 weeks of surgery

Exclusion Criteria:

* Previous thoracic surgery
* Inoperable tumor/nodule
* Unable to tolerate surgery
* History of allergies to iodides
* Breast feeding
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Visibility in situ, white light | Through study completion, an average of one year
Visibility in situ, fluorescence | Through study completion, an average of one year
Nodule malignancy | Through study completion, an average of one year

SECONDARY OUTCOMES:
Visibility ex vivo, white light | Through study completion, an average of one year
Visibility ex vivo, fluorescence | Through study completion, an average of one year

CONTACTS AND LOCATIONS:
Overall Officials: Inderpal Sarkaria, MD, Principal Investigator — University of Pittsburgh Medical Center/UPP
Locations (1):
- Department of Cardiothoracic Surgery, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No